CLINICAL TRIAL: NCT05793593
Title: FITx3 RCT: A Pilot Randomized Controlled Trial Leveraging Social Networks to Encourage Three Peers to Complete Fecal Immunochemical Testing for Colorectal Cancer
Brief Title: A Study of Using Social Networks to Encourage Three Peers to Complete Screening for Colorectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: CANCER PREVENTION FUND (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-078
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Colon Cancer Screening
Keywords: Fecal Immunochemical Testing; Screening; 23-078
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colorectal Cancer (CRC) education alone (Active Comparator): All participants will be educated, on a simplified clinical and medical background of CRC; causes and risk factors for CRC; eligibility criteria for screening; lifestyle modifications to lower risk of developing CRC; screening methods for CRC, including FIT and colonoscopy; addressing myths and misconceptions about CRC; and information about resources for low-cost and no-cost screening, screening for the uninsured and screening for those without legal immigration documentation. Participants will also be educated on elements of fecal immunochemical testing (detects signs of cancer in the stool, can be done at home and sent to a laboratory for analysis, needs to be done yearly to ensure maximal effectiveness for cancer screening). Follow-up Assessment at 8 months complete follow-up form and assist in completion of peer outreach tracker Provide reminders to encourage participants to encourage peers to get FIT tested.
  Interventions: Other: Colorectal Cancer (CRC) education alone
- FITx3 intervention and CRC education (Experimental): Provide CRC education, SN education, handouts and text message/social media posts example library. Monthly Telephone Support Provide any additional support to index participants for peer FIT testing, assist in completion of peer outreach tracker. Biweekly Text Messages. Follow-up Assessment (month 8 after intervention) Complete follow-up form and assist in completion of peer outreach tracker Provide reminders to encourage participants to encourage peers to get FIT tested.
  Interventions: Other: FITx3 intervention and CRC education

INTERVENTIONS:
Other: FITx3 intervention and CRC education — Provide CRC education, SN education, handouts and text message/social media posts example library. Monthly Telephone Support Provide any additional support to index participants for peer FIT testing, assist in completion of peer outreach tracker. Biweekly Text Messages. Follow-up Assessment (month 8 after intervention) Complete follow-up form and assist in completion of peer outreach tracker Provide reminders to encourage participants to encourage peers to get FIT tested.
  Arms: FITx3 intervention and CRC education
Other: Colorectal Cancer (CRC) education alone — CRC education alone.
  Arms: Colorectal Cancer (CRC) education alone

SUMMARY:
The Black community has higher rates of colorectal cancer and lower rates of colorectal cancer screenings than whites. Getting screened through FIT testing may help catch colorectal cancer earlier, when it is easier to treat. MSK has created a program to help people who have been FIT tested to also help their peers (family, friends, and colleagues) in their community get FIT tested. The researchers think that training people on peer outreach, such as telling people in your social network about FIT testing and how to get it, may increase the rate of colorectal cancer screening. The purpose of this study is to see if training people on peer outreach increases the number of people who get screened for colorectal cancer through FIT testing.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Black (inclusive of African, African-American, or Afro-Caribbean)
* Male
* Speaks English or French very well
* Is at least 45 years of age and no greater than 75 years of age
* Has completed FIT testing within the prior year
* Has at least 5 close network affiliates, who are Black males, and of at least 45 years of age and no greater than 75 years of age

Exclusion Criteria:

* Has a household member who has already participated (or agreed to participate)
* Has already been approached by a peer participating in the study (index participant) to complete FIT testing

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
number of people beyond the index participants who complete FIT screening | within 8 months of the index participant's enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoiral Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm